CLINICAL TRIAL: NCT03441802
Title: Gut Microbiota as a Novel Therapeutic Target for Prevention of Cardiovascular Diseases in Obese and Non-obese Adult Subjects
Brief Title: Gut Microbiota as a Therapeutic Target for CVD
Acronym: oliomicroFDG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: olio1_FDG
Record Dates: First submitted 2018-02-08; First posted 2018-02-22 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cases (Active Comparator)
  Interventions: Other: High quality extra virgin olive oil
- Controls (Other)
  Interventions: Other: High quality extra virgin olive oil

INTERVENTIONS:
Other: High quality extra virgin olive oil — Cases and controls were given 40 g/die high quality extra virgin olive oil

SUMMARY:
Background: The Mediterranean Diet (MD) is considered an healthy diet useful in the prevention of cardiovascular disease (CVD). High quality extra virgin olive oil (HQ-EVOO, [1]), an essential component of this diet, exerts a protective effect against CVD. Moreover, the gut microbiota (GM) has recently been recognized as a key factor in driving metabolic activities and involved in the stimulation of host immunity [2]. In particular, Lactic Acid Bacteria (LAB) and their probio-active cellular substances produce beneficial effects in the gastrointestinal tract, thus representing important assets in pathological conditions such as obesity and CVD [3,4].

Objective: The purpose of this study is to demonstrate that 3 months of treatment (MD with 40g/die HQ-EVOO) in 36 subjects (cases: overweight/obese vs controls: normal weight) may change their GM and inflammatory panel.

ELIGIBILITY:
Inclusion Criteria:

* normal weight subjects (M and F) with Body Mass Index (BMI) between 18.5 and 24.9 Kg/m2 following MD;
* overweight/obese subjects with a BMI ≥ 25 Kg/m2, not necessarily following MD.

Exclusion Criteria:

* eating disorders;
* recent or ongoing antibiotic therapy.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-01-08 (Actual); Primary Completion 2016-06-06 (Actual); Study Completion 2017-02-06 (Actual)

PRIMARY OUTCOMES:
anti-inflammatory cytokines | Time 0 (T0)
changes in anti-inflammatory cytokines | after 3 months from T0 (T1)

REFERENCES:
- [Background] 1) Oliveras-López M-J, Berná G, Jurado-Ruiz E, López-García de la Serrana H, Martín F. Consumption of extra-virgin olive oil rich in phenolic compounds has beneficial antioxidant effects in healthy human adults. J Funct Foods 2014;10:475-84
- [Background] 2) Hervert-Hernández D, Goñi I. Dietary Polyphenols and Human Gut Microbiota: a Review. Food Reviews International. 2011;27:154-69.
- [Background] Woting A, Blaut M. The Intestinal Microbiota in Metabolic Disease. Nutrients. 2016 Apr 6;8(4):202. doi: 10.3390/nu8040202. PMID 27058556
- [Background] Boulange CL, Neves AL, Chilloux J, Nicholson JK, Dumas ME. Impact of the gut microbiota on inflammation, obesity, and metabolic disease. Genome Med. 2016 Apr 20;8(1):42. doi: 10.1186/s13073-016-0303-2. PMID 27098727
- [Derived] Luisi MLE, Lucarini L, Biffi B, Rafanelli E, Pietramellara G, Durante M, Vidali S, Provensi G, Madiai S, Gheri CF, Masini E, Ceccherini MT. Effect of Mediterranean Diet Enriched in High Quality Extra Virgin Olive Oil on Oxidative Stress, Inflammation and Gut Microbiota in Obese and Normal Weight Adult Subjects. Front Pharmacol. 2019 Nov 15;10:1366. doi: 10.3389/fphar.2019.01366. eCollection 2019. PMID 31803056